CLINICAL TRIAL: NCT03635840
Title: The Effects of Intra Aortic Balloon Pump Prior to Revascularization on Mortality of Patients With Acute Coronary Syndrome Complicated With Cardiogenic Shock
Brief Title: The Effects of IABP Prior to Revascularization on Mortality of ACS Patients Complicated With Cardiogenic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Dafsah A. Juzar, MD, Interventional Cardiologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IABP18
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cardiogenic Shock
Keywords: IABP; Cardiogenic Shock; Myocardial Infarction
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Group of patients not receiving IABP
- Intra Aortic Balloon Pump (Experimental): Group of patients receiving Intra Aortic Balloon Pump prior to revascularization
  Interventions: Device: Intra Aortic Balloon Pump

INTERVENTIONS:
Device: Intra Aortic Balloon Pump — Intra Aortic Balloon Pump (IABP) is a circulatory mechanical support device, placed in descending aorta, distally from left subclavian artery and proximally from renal artery. IABP works with counterpulsation concept, synchronized with heart cycle. It is indicated as supportive therapy for patients undergoing revascularization, cardiogenic shock and mechanical complication.
  Balloon dilatation during dyastolic phase increasing dyastolic pressure in aorta, improving coronary vascularization and myocardial oxygen supply. In systolic phase, the balloon deflates, reducing the left ventricle afterload hence decreasing myocardial oxygen demand.
  Other Names: IABP
  Arms: Intra Aortic Balloon Pump

SUMMARY:
Prevalence of cardiogenic shock in acute coronary syndrome patients is reported at about 5-8% with high fatality. Revascularization approach has already known as the standard of care, but the usage of intra-aortic balloon pump (IABP) as mechanical circulatory support is still a controversy. IABP SHOCK II trial revealed that short-term mortality did not improved by IABP but there are several essential variabels related to mortality that are not considered in the study which are IABP initiation time and weaning protocol.This study aim to evalute the effect of IABP prior to revascularization on mortality of patients with myocardial infarction complicated with shock.

92 subjects will be enrolled in this randomized controlled trial into two groups, with and without IABP. IABP group will be receiving the intervention prior to revascularization. The primary outcomes to be sought are in-hospital and 30-day mortality after revascularization. IABP effects measured by various indicators such as Global Longitudinal Strain by echocardiography on the 1st and 3rd day, NTproBNP and ST2 level on the 1st, 3rd and 5th day, effective lactate clearance and ureum creatinine level on the 1st and 3rd day and will be compared between two groups. Continous variabel will be presented in mean ± deviation standard or median, and analized with Student's t test or Mann-Whitney U test as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Myocardial infarction patients complicated with shock
* Willing to enroll in the study (signed consent)

Exclusion Criteria:

* Age greater than 80 years old
* Heart and lung resuscitation for more than 30 minutes
* Cardiogenic shock onset >12 hours (if known) or >18 hours (if not known/patient presented in emergency department already with shock)
* Mechanical complication of myocardial infarction
* Moderate and severe aorta regurgitation
* Peripheral artery disease making IABP unfeasible
* Patients not receiving revascularization by percutaneous coronary intervention
* Patients who died before IABP insertion
* Care termination requested by family

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
30-day-Mortality | 30 days
  Mortality of patients 30 day after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dafsah Juzar, MD, Principal Investigator — National Cardiovascular Center Harapan Kita Hospital Indonesia
Locations (1):
- National Cradiovascular Center Harapan Kita Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nabel EG, Braunwald E. A tale of coronary artery disease and myocardial infarction. N Engl J Med. 2012 Jan 5;366(1):54-63. doi: 10.1056/NEJMra1112570. No abstract available. PMID 22216842
- [Background] Lindholm MG, Kober L, Boesgaard S, Torp-Pedersen C, Aldershvile J; Trandolapril Cardiac Evaluation study group. Cardiogenic shock complicating acute myocardial infarction; prognostic impact of early and late shock development. Eur Heart J. 2003 Feb;24(3):258-65. doi: 10.1016/s0195-668x(02)00429-3. PMID 12590903
- [Background] Goldberg RJ, Spencer FA, Gore JM, Lessard D, Yarzebski J. Thirty-year trends (1975 to 2005) in the magnitude of, management of, and hospital death rates associated with cardiogenic shock in patients with acute myocardial infarction: a population-based perspective. Circulation. 2009 Mar 10;119(9):1211-9. doi: 10.1161/CIRCULATIONAHA.108.814947. Epub 2009 Feb 23. PMID 19237658
- [Background] Barron HV, Every NR, Parsons LS, Angeja B, Goldberg RJ, Gore JM, Chou TM; Investigators in the National Registry of Myocardial Infarction 2. The use of intra-aortic balloon counterpulsation in patients with cardiogenic shock complicating acute myocardial infarction: data from the National Registry of Myocardial Infarction 2. Am Heart J. 2001 Jun;141(6):933-9. doi: 10.1067/mhj.2001.115295. PMID 11376306
- [Background] Acharji S, Mathur A, Lakshmanadoss U, Prasad H, Singh M, Kaluski E. Have we given up on intra-aortic balloon counterpulsation in post-myocardial infarction cardiogenic shock? Clin Cardiol. 2013 Nov;36(11):704-10. doi: 10.1002/clc.22184. Epub 2013 Sep 17. PMID 24105878
- [Background] Hochman JS, Sleeper LA, Webb JG, Dzavik V, Buller CE, Aylward P, Col J, White HD; SHOCK Investigators. Early revascularization and long-term survival in cardiogenic shock complicating acute myocardial infarction. JAMA. 2006 Jun 7;295(21):2511-5. doi: 10.1001/jama.295.21.2511. PMID 16757723
- [Background] Reynolds HR, Hochman JS. Cardiogenic shock: current concepts and improving outcomes. Circulation. 2008 Feb 5;117(5):686-97. doi: 10.1161/CIRCULATIONAHA.106.613596. No abstract available. PMID 18250279
- [Background] Werdan K, Russ M, Buerke M, Delle-Karth G, Geppert A, Schondube FA; German Cardiac Society; German Society of Intensive Care and Emergency Medicine; German Society for Thoracic and Cardiovascular Surgery; (Austrian Society of Internal and General Intensive Care Medicine; German Interdisciplinary Association of Intensive Care and Emergency Medicine; Austrian Society of Cardiology; German Society of Anaesthesiology and Intensive Care Medicine; German Society of Preventive Medicine and Rehabilitation. Cardiogenic shock due to myocardial infarction: diagnosis, monitoring and treatment: a German-Austrian S3 Guideline. Dtsch Arztebl Int. 2012 May;109(19):343-51. doi: 10.3238/arztebl.2012.0343. Epub 2012 May 11. PMID 22675405
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Jeger RV, Urban P, Harkness SM, Tseng CH, Stauffer JC, Lejemtel TH, Sleeper LA, Pfisterer ME, Hochman JS. Early revascularization is beneficial across all ages and a wide spectrum of cardiogenic shock severity: A pooled analysis of trials. Acute Card Care. 2011 Mar;13(1):14-20. doi: 10.3109/17482941.2010.538696. Epub 2011 Jan 18. PMID 21244231
- [Background] Overgaard CB, Dzavik V. Inotropes and vasopressors: review of physiology and clinical use in cardiovascular disease. Circulation. 2008 Sep 2;118(10):1047-56. doi: 10.1161/CIRCULATIONAHA.107.728840. No abstract available. PMID 18765387
- [Background] Abraham WT, Adams KF, Fonarow GC, Costanzo MR, Berkowitz RL, LeJemtel TH, Cheng ML, Wynne J; ADHERE Scientific Advisory Committee and Investigators; ADHERE Study Group. In-hospital mortality in patients with acute decompensated heart failure requiring intravenous vasoactive medications: an analysis from the Acute Decompensated Heart Failure National Registry (ADHERE). J Am Coll Cardiol. 2005 Jul 5;46(1):57-64. doi: 10.1016/j.jacc.2005.03.051. PMID 15992636
- [Background] Brodie BR, Stuckey TD, Hansen C, Muncy D. Intra-aortic balloon counterpulsation before primary percutaneous transluminal coronary angioplasty reduces catheterization laboratory events in high-risk patients with acute myocardial infarction. Am J Cardiol. 1999 Jul 1;84(1):18-23. doi: 10.1016/s0002-9149(99)00185-x. PMID 10404845
- [Background] Sjauw KD, Engstrom AE, Vis MM, van der Schaaf RJ, Baan J Jr, Koch KT, de Winter RJ, Piek JJ, Tijssen JG, Henriques JP. A systematic review and meta-analysis of intra-aortic balloon pump therapy in ST-elevation myocardial infarction: should we change the guidelines? Eur Heart J. 2009 Feb;30(4):459-68. doi: 10.1093/eurheartj/ehn602. Epub 2009 Jan 23. PMID 19168529
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Background] Fuchs RM, Brin KP, Brinker JA, Guzman PA, Heuser RR, Yin FC. Augmentation of regional coronary blood flow by intra-aortic balloon counterpulsation in patients with unstable angina. Circulation. 1983 Jul;68(1):117-23. doi: 10.1161/01.cir.68.1.117. PMID 6851038
- [Background] Abdel-Wahab M, Saad M, Kynast J, Geist V, Sherif MA, Richardt G, Toelg R. Comparison of hospital mortality with intra-aortic balloon counterpulsation insertion before versus after primary percutaneous coronary intervention for cardiogenic shock complicating acute myocardial infarction. Am J Cardiol. 2010 Apr 1;105(7):967-71. doi: 10.1016/j.amjcard.2009.11.021. Epub 2010 Feb 13. PMID 20346314
- [Background] Schwarz B, Abdel-Wahab M, Robinson DR, Richardt G. Predictors of mortality in patients with cardiogenic shock treated with primary percutaneous coronary intervention and intra-aortic balloon counterpulsation. Med Klin Intensivmed Notfmed. 2016 Nov;111(8):715-722. doi: 10.1007/s00063-015-0118-8. Epub 2015 Nov 23. PMID 26596273
- [Background] Fuernau G, Poenisch C, Eitel I, Denks D, de Waha S, Poss J, Heine GH, Desch S, Schuler G, Adams V, Werdan K, Zeymer U, Thiele H. Prognostic impact of established and novel renal function biomarkers in myocardial infarction with cardiogenic shock: A biomarker substudy of the IABP-SHOCK II-trial. Int J Cardiol. 2015 Jul 15;191:159-66. doi: 10.1016/j.ijcard.2015.04.242. Epub 2015 May 1. PMID 25965624
- [Background] Attana P, Lazzeri C, Picariello C, Dini CS, Gensini GF, Valente S. Lactate and lactate clearance in acute cardiac care patients. Eur Heart J Acute Cardiovasc Care. 2012 Jun;1(2):115-21. doi: 10.1177/2048872612451168. PMID 24062898

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT03635840/Prot_SAP_ICF_000.pdf